CLINICAL TRIAL: NCT05557994
Title: Assessment of Different Disinfection Protocols on Regenerative Potential of Mature Permanent Teeth With Necrotic Pulps Protocols
Brief Title: Assessment of Different Disinfection Protocols on Regenerative Potential of Mature Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Abanoub Raouf Ishak, Assistant lecturer, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dentistrymu
Record Dates: First submitted 2022-09-24; First posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Apical Periodontitis
MeSH Terms: conditions — Periapical Periodontitis | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood clotting (Active Comparator): Blood clotting protocol for pulp regeneration of mature teeth
  Interventions: Other: Method
- Disinfection technique (Experimental): Compare different disinfection technique
  Interventions: Other: Method

INTERVENTIONS:
Other: Method — treatment of mature teeth with apical periodontitis

SUMMARY:
Regenerative endodontic procedures have been used to successfully treat human mature permanent teeth with necrotic pulps and apical periodontitis. Many researchers have begun to apply regenerative endodontic procedures to mature teeth in adult patients. Several clinical case reports have shown complete resolution of signs and symptoms of pulp necrosis in mature teeth, even those with large periapical lesions, as well as signs of pulp canal obliteration. The aim of this study is to assess the regenerative potential of mature permanent teethwith necrotic pulps after disinfecting the root canal using diode laser andcompare it with dynamic agitation of xp-endo finisher and conventionaltriple antibiotic paste

ELIGIBILITY:
Inclusion Criteria:

Patients with mature teeth. Patients with periapical periodontitis. Maxillary anterior teeth only will be involved. Patients should be free from any systemic disease that may affect normal healing and predictable outcome.

Patients who will agree to the consent and will commit to follow up period.

Exclusion Criteria:

* Patients with immature roots. - Immuno-compromised patients, including patients who self-reportedto be a carrier of HIV, hepatitis, undergoing steroid therapy, thosewho self-reported with genetic or systemic diseases that could resultin a reduced immune response.- All patients who respond positive to allergic patch test [tripleantibiotic paste] and drugs.- Pregnant and lactating women.- Patients who could/would not participate in a 1-year follow-up.- Teeth with previous endodontic therapy performed. - Teeth with periodontal involvement. - Teeth with calcified canals.- Presence of external or internal root resorption.- Teeth with root fractures (checked with pre-operative radiographsusing horizontal and vertical angulations)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Clinical success | 9 months
  pulp vitality testing using electric pulp tester which detect response of pulp to electric current

SECONDARY OUTCOMES:
Radiographic success | 9 months
  healing of apical periodontitis by detecting change in apical radiolucency and absences of apical bone resorption

CONTACTS AND LOCATIONS:
Locations (1):
- Abanoub Raouf, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No